CLINICAL TRIAL: NCT04620980
Title: Assessing the Polygenic Burden of Rare Disruptive Mutations in Parkinson's Disease: a Novel Diagnostic Test to Predict Parkinson's Disease Risk
Brief Title: Assessing the Polygenic Burden of Rare Disruptive Mutations in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Teresa Esposito, Head of CNR Unit, Neuromed IRCCS
Other Study IDs: RF-2019-12370224
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples for purification of DNA, RNA, plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants will be assessed for disease progression: Hoehn and Yahr stadium, MDS-UPDRS part III, MoCA test, no motor symptoms, therapy and LID occurrence.
  Participants will be subjected to peripheral blood sampling for the purification of DNA, RNA, plasma and serum.
  DNA of each participant will be analysed by targeted resequencing of a disease-specific gene panel including about 100 genes related to Parkinson's Disease, autophagy and levodopa induced Dyskinesia (LID).
  Interventions: Diagnostic Test: targeted resequencing
- controls: Participants will be assessed for the presence of disease. Participants will be subjected to peripheral blood sampling for the purification of DNA, RNA, plasma and serum.
  DNA of each participant will be analysed by targeted resequencing of a disease-specific gene panel including about 100 genes related to Parkinson's Disease, autophagy and levodopa induced Dyskinesia (LID).
  Interventions: Diagnostic Test: targeted resequencing

INTERVENTIONS:
Diagnostic Test: targeted resequencing — The investigators will use a disease-specific gene panel including about 100 genes related to Parkinson's Disease, autophagy and levodopa induced Dyskinesia (LID).

SUMMARY:
The project intends to assess the polygenic burden of rare disruptive mutations in Parkinson's disease (PD) and how they influence the phenotype/pathological heterogeneity of disease.

DETAILED DESCRIPTION:
The investigators intend to extend the genetic analysis to a cohort of 300 PD cases and 300 healthy subjects (wife / husband of the patients) that will be recruited at Scientific Institute for Research, Hospitalization and Healthcare (IRCCS) Neuromed.

After signed informed consent patients will be assessed for disease progression (Hoehn and Yahr stadium, Movement Disorder Society-Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS), Montreal Cognitive Assessment (MoCA) test, no motor symptoms, therapy and levodopa induced Dyskinesia (LID) occurrence). Each patient and control will be subjected to peripheral blood sampling for the isolation of DNA, RNA, plasma and serum. The investigators will use a disease-specific gene panel including about 100 genes related to Parkinson's Disease, autophagy and levodopa induced Dyskinesia (LID).

Bioinformatics analysis will allow to catalog in a database the identified variants/mutations according to their frequency and characteristics.

The investigators will specifically assess if the inheritance of multiple rare deleterious variants in Parkinson's Disease genes is predictive of disease risk.

The presence of one or more variants will be tested for association with phenotypic manifestation of Parkinson's Disease (motor, non-motor, and cognitive signs, as well as age at onset, LID and neuroimaging changes) to assess the variant burden effect on progression, and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two out the following cardinal signs: resting tremor, cogwheel rigidity, bradykinesia, asymmetrical onset of symptoms and symptomatic response to L-dopa (levodopa).

Exclusion Criteria:

* Previous thalamotomy on the implanted sides;
* Significant brain atrophy or structural damage seen on CT or MRI;
* Marked cognitive dysfunction;
* Active psychiatric symptoms;
* Concurrent neurological disorders;
* Other uncontrolled medical disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes 300 PD patients and 300 age/gender-matched controls. All PD patients will be diagnosed at the IRCCS Neuromed and followed-up (at least for 3 years) for disease progression.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of PD patients and controls | three years
  disease progression (Hoehn and Yahr stadium, MDS-UPDRS part III, MoCA test, no motor symptoms, therapy and LID occurrence
identification of variants/mutations | two years
  assessing if the inheritance of multiple rare deleterious variants in PD genes is predictive of PD risk.
association with phenotypic manifestation of PD | three years
  The presence of one or more variants will be tested for association with phenotypic manifestation of PD (motor, non-motor, and cognitive signs, as well as age at onset, LID and neuroimaging changes) to assess the variant burden effect on progression, and prognosis of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Esposito, PhD, Principal Investigator — Head of CNR Unit
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
genetics data